CLINICAL TRIAL: NCT06900933
Title: Reconstruction of Horizontally Deficient Atrophic Maxillary Ridges Using Retromolar Blocks With and Without Coverage Using Collagen Membrane (Randomized Clinical Trials)
Brief Title: Reconstruction of Deficient Maxillary Ridges Using Retromolar Blocks With and Without Collagen Membrane
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohannad Ahmed Ismail, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0-0002-9582-5106
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Bone Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group A: Retromolar bone block covered with collagen membrane. (Experimental): The onlay bone block harvested from retromolar region and fixed with micro screws, a mixture of autogenous and xenogenic particulate bone graft is going to be packed in between the bone block and recipient site. The assembly is going to be covered with native collagen membrane and fixed with titanium bone tacks.
  Interventions: Procedure: Onlay bone block covered with collagen membrane
- Control Group B: Retromolar bone block without collagen membrane. (Active Comparator): The onlay bone block harvested from retromolar region and fixed with micro screws, a mixture of autogenous and xenogenic particulate bone graft is going to be packed in between the bone block and recipient site.
  Interventions: Procedure: Onlay bone block without collagen membrane

INTERVENTIONS:
Procedure: Onlay bone block covered with collagen membrane — Onlay bone block covered with collagen membrane
  Arms: Study Group A: Retromolar bone block covered with collagen membrane.
Procedure: Onlay bone block without collagen membrane — Onlay bone block covered without collagen membrane
  Arms: Control Group B: Retromolar bone block without collagen membrane.

SUMMARY:
Is the use of collagen membrane on top of particulate bone mixture covered by onlay bone block in Maxilla better than the use of mixture of particulate bone covered by onlay bone block without the use of collagen membrane, in terms of bone quantity?

DETAILED DESCRIPTION:
Soft tissue dehiscence could result due to flap irritation as a result of, closure under tension, intraoperative or postoperative recipient site infection, postoperative edema, which in turns compromises stability of onlay bone blocks thus osseintegration of bone block. Any attempt of bone recontouring and resuturing fails since there is no vascular bed. Ideal requirements of barrier membranes are, they should be biological compatible, they must act as a barrier membrane, unwanted fibroblasts should be hindered from entrance while allowing diffusion of nutrients, tissue integration (biological adhesion), tissues should be able to grow into the membrane but not through it. Space maintainer, it should be sufficiently stiff, so as not to collapse into the underlying particulate bone under the pressure of soft tissue and it should be ease in its manipulation, adaptation and handling, as for example, collagen membrane. Some types of collagen membrane, contain some degrees of stretchability example Geistlich Bio-Gide or Jason Membrane Botiss.

ELIGIBILITY:
Inclusion Criteria:

* Patients with maxillary residual alveolar bone height not less than 8 mm.
* Alveolar bone width from less than or equal 5 mm.
* Both genders.
* At least missing single tooth.
* Previous Failed Implants.
* Previous Failed Grafting.

Exclusion Criteria:

* • Heavy smokers more than 20 cigarettes per day.

  * Patients with alcohol abuse
  * Patients with narcotic abuse.
  * Patients with bone disease that may affect normal healing, example; hyperparathyroidism.
  * Patients had radiotherapy and chemotherapy in head and neck.
  * Patients had neoplasms in sites to be grafted.
  * Patients with Metabolic diseases uncontrolled diabetic patients, Glycated hemoglobin (Hb A1c) more than 7 mg\dl.
  * Pregnant females.
  * Patients with Para functional habits, apprehensive and non-cooperative.
  * Bone pathology related to the site to be grafted.
  * Psychological problems, stress situation (socially or professionally), emotional instability, and unrealistic patients' expectations.
  * Intraoral soft and hard tissue pathology.
  * Systemic condition that contraindicate implant placement.
  * Under the age of 18 years.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Quantity of bone gain. | At 5 months from ridge augmentation.
  Measured using linear measurements from Cone Beam Computed Tomography in millimeters.

SECONDARY OUTCOMES:
Soft Tissue Dehiscence | Baseline 1st Week. Written Binary Numerical Yes or No.
  Exposure of bone block assembly and impaired healing

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammerle CH, Jung RE. Bone augmentation by means of barrier membranes. Periodontol 2000. 2003;33:36-53. doi: 10.1046/j.0906-6713.2003.03304.x. No abstract available. PMID 12950840
- [Background] Cash and Alex: 20 years of guided bone regeneration in implant dentistry, 2nd ed. (2009).
- [Background] Urban, I A., Nagrusky H, Lozada JM:
- [Background] Urban, I A., Nagrusky H, Lozada JM.:
- [Background] Pellegrino G, Lizio G, Corinaldesi G, Marchetti C. Titanium Mesh Technique in Rehabilitation of Totally Edentulous Atrophic Maxillae: A Retrospective Case Series. J Periodontol. 2016 May;87(5):519-28. doi: 10.1902/jop.2016.150432. Epub 2016 Jan 12. PMID 26759078
- [Background] Polis-Yanes C, Cadenas-Sebastian C, Gual-Vaques P, Ayuso-Montero R, Mari-Roig A, Lopez-Lopez J. Guided Bone Regeneration of an Atrophic Maxilla Using Heterologous Cortical Lamina. Case Rep Dent. 2019 Jun 11;2019:5216362. doi: 10.1155/2019/5216362. eCollection 2019. PMID 31308978
- [Background] Jensen J, Sindet-Pedersen S. Autogenous mandibular bone grafts and osseointegrated implants for reconstruction of the severely atrophied maxilla: a preliminary report. J Oral Maxillofac Surg. 1991 Dec;49(12):1277-87. doi: 10.1016/0278-2391(91)90303-4. PMID 1955919
- [Background] Montazem A, Valauri DV, St-Hilaire H, Buchbinder D. The mandibular symphysis as a donor site in maxillofacial bone grafting: a quantitative anatomic study. J Oral Maxillofac Surg. 2000 Dec;58(12):1368-71. doi: 10.1053/joms.2000.18268. PMID 11117684